CLINICAL TRIAL: NCT07055126
Title: Nutritional Resources and Techniques to Enhance the Diets of Young Children
Brief Title: Nutritional Resources and Techniques for Young Children
Acronym: NURTURE-Diet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Elaine McCarthy, Principal Investigator, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ECM 4 (g) 02/07/2024
Record Dates: First submitted 2025-05-29; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Healthy
Keywords: young children; nutrition education; dietary assessment; nutritional resources

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Parents/guardians of study participants will be provided with basic healthy eating advice, as per the Food Safety Authority of Ireland's Food-Based Dietary Guidelines for 1-5-year-olds (Food Safety Authority of Ireland, 2020).
- Intervention Group (Experimental): Parents/guardians of study participants will be given individualised dietary counselling, coaching and resource provision around healthy eating, with a particular focus on incorporating fresh meat and vegetables into a healthy, sustainable and safe diet for young children.
  Interventions: Other: Individualised dietary counselling, coaching and resource provision around healthy eating for young children

INTERVENTIONS:
Other: Individualised dietary counselling, coaching and resource provision around healthy eating for young children — Study participants randomised to receive the intervention will receive nutrition education support, through individualised dietary counselling, coaching and resource provision around healthy eating, with a particular focus on incorporating fresh meat and vegetables into a healthy, sustainable and safe diet for young children. Those in the control group will not receive this individualised nutrition education and supports.
  Arms: Intervention Group

SUMMARY:
This randomised controlled dietary intervention study aims to test the effect of introducing fresh meat and vegetable-based recipes and targeted dietary resources into a healthy, sustainable toddler diet on dietary intakes relative to a control group consuming a standard diet based on Irish healthy eating guidelines.

This study aims to recruit 80 young children (24-42 months old) who will be randomised to an intervention (provided with individualised dietary counselling, alongside a targeted healthy eating resource, focused on incorporating fresh red meat and vegetable based recipes into a sustainable and safe diet for young children), or control group receiving (provided with basic healthy eating advice as per the Food Safety Authority of Ireland's Food-Based Dietary Guidelines for 1-5-year-olds).

Participants will:

* Include any of the recipes in their child's diet on 3 occasions during the week, for 12 weeks
* Complete a variety of validated nutrition and feeding questionnaires
* Complete 2 onsite visits, at the baseline and endpoint of the intervention period

The provision of targeted dietary counselling with nutritional resources and techniques will allow us to investigate the impact of these strategies on improving the overall diet of young children.

ELIGIBILITY:
Inclusion Criteria:

* Child aged between 24-42 months (at time of study recruitment).
* In general good health.
* Following an unrestricted diet.
* Capable of completing the study assessments.
* Parent/guardian must be willing to provide written informed consent for their child's participation.

Exclusion Criteria:

- Follows a vegetarian or vegan or meat-avoidant diet.

Ages: 24 Months to 42 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in dietary intake of key nutrients (iron, zinc, vitamin A, vitamin B12, protein and total energy) from baseline to 12 weeks | From baseline to 12 weeks
  Assessment of change in dietary intake of iron, zinc, vitamin A, vitamin B12, protein, and total energy from baseline to week 12 in toddlers (aged 24-42 months), as measured by a 2-day weighed food and drink diary analyzed using Nutritics software.

SECONDARY OUTCOMES:
Change in weight (kilograms) from baseline to 12 weeks | From baseline to 12 weeks
  Measured in kilograms using calibrated weighing scales
Change in height (meters) from baseline to 12 weeks | From baseline to 12 weeks
  Measured in meters using a stadiometer following standardised procedures
Parent reported feasibility and acceptability of the healthy eating resource and recipes | Week 12 (Endpoint Visit)
  A 20-item self-administered questionnaire developed for this study to evaluate the feasibility and acceptability of healthy eating resources and trial recipes provided as part of the NURTURE-Diet intervention.
  The questionnaire assesses parental experiences with recipe preparation (including ease, clarity of instructions, required time, and availability of kitchen equipment) through open-ended questions and Likert-scale questions. Child and family acceptability of the recipes (including taste, texture, aroma, appearance, and overall acceptance) is measured using a 5-point Likert scale. The questionnaire is administered at the participant's endpoint visit (week 12).
Change in mean parental food neophobia score as measured by the Food Neophobia Scale from baseline to 12 weeks | From baseline to 12 weeks
  The Food Neophobia Scale (FNS) is a validated self-administered questionnaire that assesses an individual's reluctance to consume novel or unfamiliar foods. The food neophobia scale is used to assess levels of food neophobia among adults.
  The scale includes 10 items rated on a 7 point likert scale (1=Strongly disagree, 7= Strongly agree). Five items are reverse scored.
  After reverse scoring is applied, the 10 items are summed to produce a total score (minimum=10, maximum =70). Higher scores indicate greater food neophobia, characterized by a strong avoidance or refusal of unfamiliar foods (i.e., a worse outcome).
Change in mean score on the Cooking Skills Questionnaire (CSQ) from baseline to 12 weeks | From baseline to 12 weeks
  The Cooking Skills Questionnaire (CSQ) is a validated self-administered questionnaire measure assessing parents' confidence in performing a range of cooking skills, such as chopping, baking, stir-frying, steaming, and following recipes. The cooking skills questionnaire includes 14 items, each rated on a 7-point Likert scale (1 = Very poor, 7 = Very good).
  Items are averaged to produce a mean score (Minimum = 1, Maximum = 7). Higher scores reflect greater confidence in cooking skills, which is considered a positive outcome in the context of this intervention.
Change in mean score on the Food Skills Questionnaire (FSQ) from baseline to 12 weeks | From baseline to 12 weeks
  The food skills questionnaire (FSQ) is a validated self-report measure that assesses parents' confidence in practical food-related skills, including meal planning, budgeting, food label use, and using leftovers. The food skills questionnaire consists of 19 items, each rated on a 7-point Likert scale (1 = Very poor, 7 = Very good).
  Items are averaged to produce a mean score (Minimum = 1, Maximum = 7). Higher scores indicate greater confidence and frequency in using food-related skills, which is considered a positive outcome in the context of this intervention.
Change in frequency of parental inclusion of children in meal preparation and cooking activities from baseline to 12 weeks | From baseline to 12 weeks
  Parental behavior related to involving children in food preparation and cooking activities will be assessed using two validated self-report items.
  Each item is rated on a 6-point frequency scale:
  1 = Never, 2 = Less than once a week, 3 = Once a week, 4 = Several times a week, 5 = Most days, 6 = Every day.
  Responses will be averaged to calculate a mean score for each participant. Minimum = 1, Maximum = 6.
  Higher scores indicate more frequent inclusion of children in food-related activities, which is considered a positive outcome in the context of this intervention.
Change in mean score on the Perceived Responsibility subscale of the Child Feeding Questionnaire (CFQ) from baseline to 12 weeks | From baseline to 12 weeks
  The Child Feeding Questionnaire is a validated self reported assessment of parental feeding practice. The Perceived Responsibility subscale assesses the extent to which parents believe they are responsible for deciding their child's food intake. It includes 3 items, each rated on a 5-point Likert scale (1 = Never, 5 = Always).
  Items in the perceived responsibility sub-scale are combined to create a mean score. (Minimum = 1, Maximum = 5). Higher scores indicate greater perceived parental responsibility for their child's diet (i.e., a better outcome).
Change in mean score on the Perceived Parent Weight subscale of the Child Feeding Questionnaire (CFQ) from baseline to 12 weeks | From baseline to 12 weeks
  The Child Feeding Questionnaire is a validated self reported assessment of parental feeding practice. The Perceived Parent Weight subscale evaluates how parents perceive their own weight status. This scale includes 4 items, each rated on a 5-point Likert scale (1 = Markedly Underweight, 5 = Markedly Overweight).
  Items in the Perceived Parent Weight sub-scale are combined to create a mean score. (Minimum = 1, Maximum = 5).Higher scores indicate increased self-perception of being overweight. Values approaching the minimum or maximum of the scale represent less desirable outcomes.
Change in mean score on the Perceived Child Weight subscale of the Child Feeding Questionnaire (CFQ) from baseline to 12 weeks | From baseline to 12 weeks
  The Child Feeding Questionnaire is a validated self reported assessment of parental feeding practice. The Perceived Child Weight subscale evaluates how parents perceive their child's weight status. This scale includes 3 items, each rated on a 5-point Likert scale (1 = Noticeably Underweight, 5 = Noticeably Overweight).
  Items in the Perceived Child Weight sub-scale are combined to create a mean score. (Minimum = 1, Maximum = 5).Higher scores indicate that parents percieve their child to be heavier. Values approaching the minimum or maximum of the scale represent less desirable outcomes.
Change in mean score on the Concern about Child Weight subscale of the Child Feeding Questionnaire (CFQ) from baseline to 12 weeks | From baseline to 12 weeks
  The Child Feeding Questionnaire is a validated self reported assessment of parental feeding practice. The Concern about Child Weight subscale measures parental concern about their child becoming overweight. This scale includes 3 items, each rated on a 5-point Likert scale (1 = Unconcerned, 5 = Concerned).
  Items in the concern about child weight sub-scale are combined to create a mean score. (Minimum = 1, Maximum = 5).Higher scores indicate greater concern about the child's weight, which may reflect the percieved risk of the child becoming overweight or an overly controling feeding approach (i.e, a worse outcome).
Change in mean score on the Restriction subscale of the Child Feeding Questionnaire (CFQ) from baseline to 12 weeks | From baseline to 12 weeks
  The Child Feeding Questionnaire is a validated self reported assessment of parental feeding practice. The restriction subscale measures the extent to which parents restrict their child's access to certain foods. This scale includes 8 items, each rated on a 5-point Likert scale (1 = Disagree, 5 = Agree).
  Items in the restriction sub-scale are combined to create a mean score. (Minimum = 1, Maximum = 5). Higher scores indicate greater use of restrictive feeding practices and may be considered a worse outcome.
Change in mean score on the pressure to eat subscale of the Child Feeding Questionnaire (CFQ) from baseline to 12 weeks | From baseline to 12 weeks
  The Child Feeding Questionnaire is a validated self reported assessment of parental feeding practice. The pressure to eat subscale measures the extent to which parents pressure their child to eat more food. This scale includes 4 items, each rated on a 5-point Likert scale (1 = Disagree, 5 = Agree).
  Items in the restriction sub-scale are combined to create a mean score. (Minimum = 1, Maximum = 5). Higher scores indicate greater exertion of pressure on children to eat more food despite hunger or satiety cues (i.e., a worse outcome).
Change in mean score on the Monitoring subscale from the Child Feeding Questionnaire (CFQ) from baseline to 12 weeks | From baseline to 12 weeks
  The Child Feeding Questionnaire is a validated self reported assessment of parental feeding practice. The monitoring subscale measures the extent to which parents monitor the foods that their child eats. This scale includes 3 items, each rated on a 5-point Likert scale (1 = Disagree, 5 = Agree).
  Items in the monitoring sub-scale are combined to create a mean score. (Minimum = 1, Maximum = 5). Higher scores indicate greater monitoring of childrens dietary intakes, often considered to be a positive outcome.
Change in mean score on the Food Responsiveness subscale of the Child Eating Behaviour Questionnaire (CEBQ) from baseline to 12 weeks | From baseline to 12 weeks
  The Child Eating Behaviour Questionnaire (CEBQ) is a validated parent-reported measure assessing children's eating behaviours. The food responsiveness sub scale consists of items rated on a 5-point Likert scale ( 1=Never, 5= Always).
  Items in the food responsiveness sub-scale are combined to create a mean score. Minimum =1, Maximum = 5. Higher scores indicate greater food responsiveness, reflecting increased appetite and tendency to eat in response to external food cues (i.e, a worse outcome).
Change in mean score on the Emotional Overeating subscale of the Child Eating Behaviour Questionnaire (CEBQ) from baseline to 12 weeks | From baseline to 12 weeks
  The Child Eating Behaviour Questionnaire (CEBQ) is a validated parent-reported measure assessing children's eating behaviours. The emotional overeating sub scale consists of items rated on a 5-point Likert scale ( 1=Never, 5= Always).
  Items in the emotional overeating sub-scale are combined to create a mean score. Minimum =1, Maximum = 5. Higher scores indicate greater emotional overeating, characterized by children eating more in response to negative emotions (i.e, a worse outcome).
Change in mean score on the Enjoyment of Food subscale of the Child Eating Behaviour Questionnaire (CEBQ) from baseline to 12 weeks | From baseline to 12 weeks
  The Child Eating Behaviour Questionnaire (CEBQ) is a validated parent-reported measure assessing children's eating behaviours. The enjoyment of food sub scale consists of items rated on a 5-point Likert scale ( 1=Never, 5= Always).
  Items in the enjoyment of food sub-scale are combined to create a mean score. Minimum =1, Maximum = 5. Higher scores indicate enjoyment of food, characterized by children displaying more interest in eating. Scores closer to the minimum or maximum values of the scale suggest undesirable eating behaviour.
Change in mean score on the Desire to Drink sub-scale of the Child Eating Behaviour Questionnaire (CEBQ) from baseline to 12 weeks | From baseline to 12 weeks
  The Child Eating Behaviour Questionnaire (CEBQ) is a validated parent-reported measure assessing children's eating behaviours. The desire to drink sub-scale consists of items rated on a 5-point Likert scale ( 1=Never, 5= Always).
  Items in the desire to drink sub-scale are combined to create a mean score. Minimum =1, Maximum = 5. Higher scores indicate a greater desire to drink, often reflecting behaviours such as increased sugary beverage consumption and drinking without hunger cues (i.e., a worse outcome)
Change in mean score on the Satiety Responsiveness sub-scale of the Child Eating Behaviour Questionnaire (CEBQ) from baseline to 12 weeks | From baseline to 12 weeks
  The Child Eating Behaviour Questionnaire (CEBQ) is a validated parent-reported measure assessing children's eating behaviours. The satiety responsiveness sub-scale consists of items rated on a 5-point Likert scale (1=Never, 5= Always), with some items reverse scored.
  Items in the satiety responsiveness sub-scale are combined, after applying reverse scoring, to create a mean score. Minimum =1, Maximum = 5. Higher scores indicate greater satiety responsiveness, reflecting the ability to stop eating when full (i.e., a better outcome).
Change in mean score on the Slowness in Eating sub-scale of the Child Eating Behaviour Questionnaire (CEBQ) from baseline to 12 weeks | From baseline to 12 weeks
  The Child Eating Behaviour Questionnaire (CEBQ) is a validated parent-reported measure assessing children's eating behaviours. The slowness in eating sub-scale consists of items rated on a 5-point Likert scale (1=Never, 5= Always), with some items reverse scored.
  Items in the slowness in eating sub-scale are combined, after applying reverse scoring, to create a mean score. Minimum =1, Maximum = 5. Higher scores indicate slower eating pace, with values closer to the minimum or maximum of the scale suggesting atypical eating behaviour
Change in mean score on the Emotional Undereating sub-scale of the Child Eating Behaviour Questionnaire (CEBQ) from baseline to 12 weeks | From baseline to 12 weeks
  The Child Eating Behaviour Questionnaire (CEBQ) is a validated parent-reported measure assessing children's eating behaviours. The emotional undereating sub-scale consists of items rated on a 5-point Likert scale (1=Never, 5= Always).
  Items in the emotional undereating sub-scale are combined to create a mean score. Minimum =1, Maximum = 5. Higher scores indicate greater emotional undereating, characterized by reduced food intake in response to negative emotions (i.e., a worse outcome).
Change in mean score on the Food Fussiness sub-scale of the Child Eating Behaviour Questionnaire (CEBQ) from baseline to 12 weeks | From baseline to 12 weeks
  The Child Eating Behaviour Questionnaire (CEBQ) is a validated parent-reported measure assessing children's eating behaviours. The food fussiness sub-scale consists of items rated on a 5-point Likert scale (1=Never, 5= Always), with some items reverse scored.
  Items in the food fussiness sub-scale are combined, after applying reverse scoring, to create a mean score. Minimum =1, Maximum = 5. Higher scores indicate greater food fussiness, characterized by picky eating and a refusal to eat novel foods (i.e., a worse outcome).

CONTACTS AND LOCATIONS:
Locations (2):
- Ireland (2):
  - Human Nutrition Studies Unit, Cork, Cork
  - Human Nutrition Studies Unit, School of Food and Nutritional Sciences, University College Cork., Cork, Ireland

IPD SHARING:
Plan to Share IPD: No